CLINICAL TRIAL: NCT07285395
Title: A Phase I Investigator-Initiated Trial (IIT) of AT1019 Combined With Stereotactic Body Radiation Therapy (SBRT) and PD-1 Inhibitor for Advanced Solid Tumors
Brief Title: AT1019 Plus SBRT and PD-1 Inhibitor for Advanced Solid Tumors: An IIT Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT1019-01
Record Dates: First submitted 2025-11-19; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AT1019+SBRT+PD-1 inhibitor (Experimental)
  Interventions: Drug: AT1019

INTERVENTIONS:
Drug: AT1019 — 1. First receive PD-1 inhibitor treatment.
  2. Undergo SBRT, which will be given in 3 to 5 fractions, with each fraction ranging from 6Gy to 18Gy, and the treatment will be administered once a week.
  3. Receive intratumoral injection of AT1019 within 1 to 2 days after each SBRT session.
  Other Names: PD-1 inhibitor; SBRT

SUMMARY:
The goal of this clinical trial is to assess the safety and tolerability of AT1019 when used in combination with SBRT and PD-1 inhibitor, and determine the maximum tolerated dose (MTD) of AT1019 in the combination therapy of SBRT and PD-1 inhibitor in patients with advanced solid tumors. The main questions it aims to answer are:

Is the combination of AT1019, SBRT and PD-1 inhibitor safe and well-tolerated in patients with advanced solid tumors? What is the maximum tolerated dose (MTD) of AT1019 when combined with SBRT and PD-1 targeted immunotherapy?

Participants will:

* First receive PD-1 inhibitor treatment as scheduled.
* Undergo SBRT, which will be given in 3 to 5 fractions, with each fraction ranging from 6Gy to 18Gy, and the treatment will be administered once a week.
* Receive intratumoral injection of AT1019 within 1 to 2 days after each SBRT session.
* Undergo imaging examinations every 6 weeks (with a tolerance of ±1 week) to evaluate the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 years.
2. Signed the informed consent form and have the psychological capacity to understand it.
3. Patients with advanced solid malignant tumors (such as non-small cell lung cancer, renal cell carcinoma, head and neck cancer, cervical cancer, and urothelial carcinoma) who are receiving immunotherapy and planned to undergo SBRT. Patients are eligible if they achieved at least stable disease during previous immunotherapy.
4. Patients' disease must be evaluated according to RECIST v.1.1.
5. Presence of metastatic lesions amenable to radiation therapy.
6. Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 1.
7. No evidence of clinically significant conduction abnormalities or active ischemia on electrocardiogram (ECG), as judged by the investigator.
8. Acceptable organ and bone marrow function as demonstrated by the following criteria:

(1) Absolute neutrophil count > 1500 cells/μL; (2) Platelet count > 50,000 cells/μL; (3) Total bilirubin ≤ 1.5 times the upper limit of normal (ULN); (4) Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 times the ULN; if hepatic metastasis exists, AST/ALT < 5 times the ULN; (5) Serum creatinine < 1.5 mg/dL and creatinine clearance ≥ 50 mL/min as calculated by the Cockcroft-Gault formula; (6) Prothrombin time (PT)/partial thromboplastin time (PTT) ≤ 1.5 times the ULN.

9. Females of childbearing potential (defined as those who have experienced menarche and have not undergone successful surgical sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or are not postmenopausal (defined as at least 12 months of amenorrhea with appropriate clinical documentation, such as age > 45 years)) must undergo a serum pregnancy test prior to the first administration of study treatment and confirm a negative result.

10. Male and female patients of childbearing potential must agree to use two effective contraceptive methods throughout the study period.

Exclusion Criteria:

1. Previous therapeutic radiotherapy to the same lesion.
2. Failure to recover to grade 1 or lower from clinically significant adverse events related to prior anticancer therapy, as judged by the investigator.
3. Previous grade 4 toxicity attributed to immunotherapy.
4. Known untreated brain metastases or treated but unstabilized brain metastases (central nervous system lesions shown on scan to be non-progressive and not requiring corticosteroid use) ≥ 4 weeks prior to enrollment.
5. QT/QTc interval prolongation (QTc interval > 470 milliseconds).
6. Uncontrolled intercurrent illnesses (including but not limited to ongoing or active infections, symptomatic congestive heart failure, unstable angina, arrhythmias, or psychiatric/social conditions) that, in the investigator's judgment, would limit the patient's compliance with study requirements.
7. Pregnant or lactating women.
8. The Sponsor reserves the right to exclude any patient based on pre-study medical history, physical examination findings, clinical laboratory results, prior medications, or other enrollment criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Four weeks after the end of the combination therapy.
  Determine the DLT of AT1019 in the combination therapy of SBRT and PD-1 inhibitor.
Maximum tolerated dose (MTD) | Four weeks after the end of the combination therapy.
  Determine the MTD of AT1019 in the combination therapy of SBRT and PD-1 inhibitor.
Adverse event (AE) | From the first dose to 12 months after the last dose.
  Rates and severity of AEs assessed by CTCAE v5.0 criterion.

SECONDARY OUTCOMES:
Abscopal effect rate | 3 months after the end of the combination therapy.
  The proportion of patients with an abscopal response assessed by RECIST v1.1 criterion.
Objective response rate (ORR) | Six weeks (with a tolerance of ±1 week) after the end of the combination therapy.
  To evaluate ORR of AT1019 in combination with SBRT and PD-1 inhibitor based on RECIST v1.1 criterion.
Disease control rate (DCR) | Six weeks (with a tolerance of ±1 week) after the end of the combination therapy.
  To evaluate DCR of AT1019 in combination with SBRT and PD-1 inhibitor based on RECIST v1.1 criterion.
Progress-free survival (PFS) | 5 years after the end of the combination therapy.
  To evaluate PFS of AT1019 in combination with SBRT and PD-1 inhibitor. PFS was defined from date of recruit to date of first documentation of progression or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No